CLINICAL TRIAL: NCT06132035
Title: Phase I Clinical Study to Evaluate the Safety of CG-P5 Peptide Eye Drops (Self-administered and Topically Applied) in Patients Diagnosed With Age-related Wet Macular Degeneration
Brief Title: Study to Evaluate the Safety of CG-P5 Peptide Eye Drops in Patients Diagnosed With Age-related Wet Macular Degeneration
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Caregen Co. Ltd. (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CG_P5_2023W1
Record Dates: First submitted 2023-10-24; First posted 2023-11-15 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Age-related Wet Macular Degeneration
Keywords: Age-Related Macular Degeneration; Macular Degeneration; wAMD
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CG-P5 peptide eye drops (Experimental)
  Interventions: Drug: CG-P5 peptide
- Placebo Eye drops (Placebo Comparator)
  Interventions: Drug: Placebo
- Intravitreal injection of Eylea® (Active Comparator)
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: CG-P5 peptide — Patient will instill daily 1 package of CG-P5 peptide eye drops in the study eye [self-administered] using the single use tear-off disposable packaging
  Arms: CG-P5 peptide eye drops
Drug: Placebo — Patient will instill daily 1 package of Placebo eye drops in the study eye [self-administered] using the single use tear-off disposable packaging
  Arms: Placebo Eye drops
Drug: Aflibercept Injection [Eylea] — Patient will receiver Eylea® (Aflibercept) intravitreal injection once in a month
  Arms: Intravitreal injection of Eylea®

SUMMARY:
This will be a randomized, comparative, parallel, clinical study to assess initial safety and tolerability of CG-P5 peptide eye drops compared to placebo in patients diagnosed with age-related wet macular degeneration

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥50 years of age
* Willing and able to provide written informed consent
* Diagnosis of age-related wet macular degeneration (wAMD) in the study eye as determined by the investigator on fundus examination
* Primary or recurrent active choroidal neovascularization (CNV) lesions involving the foveal center secondary to age-related wet macular degeneration in any one of the eyes. (If both eyes are affected and eligible, the eye with the worse BCVA, as assessed at screening, will be selected as the study eye
* Best corrected visual acuity (BCVA) of 75-25 eye Early Treatment of Diabetic Retinopathy Study (ETDRS) letters (approximate Snellen equivalent between 20/ 32 to 20/320) inclusive before pupil dilation assessed at the initial testing distance of 4 meters
* Central Subfield Thickness (CST thickness) ≥ 250 microns on SD-OCT (exclusive of subretinal pigment epithelial fluid, inclusive of SRF)
* Presence of SRF and/or IRF on SD-OCT
* Total lesion size not greater than 12 disc areas (30.48 mm2) (1 disc area = 2.54 mm2) on FA
* If present, subretinal hemorrhage must comprise < 50% of the total lesion area on FA, SD-OCT, or FAF
* No subfoveal fibrosis or atrophy on FA, SD-OCT, or FAF
* Active CNV membranes with subfoveal leakage or juxtafoveal leakage too close for laser photocoagulation
* Females who are of non-childbearing potential (surgically sterile or menopausal) OR if of childbearing potential using effective birth control and non-pregnant & non-lactating
* Ability to follow protocol requirements

Exclusion Criteria:

* Patients having additional eye disease in the posterior segment of study eye other than wAMD
* Any other pathology involving the CNV lesion like retro foveolar atrophy or permanent structural damage to fovea or fibrosis/ hemorrhage involving fovea > 50 % of lesion area of study eye that can affect the efficacy of drug
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment, retinal pigment epithelial tear involving the macula or macular hole (stage 3 or 4) in the study eye
* Aphakia or absence of the posterior capsule in the study eye
* History or expectation of the following surgery in the study eye:

  * Vitrectomy within last 1 month
  * Cataract surgery or Lasik within the last 3 months
  * Planned cataract removal surgery during the study
* A history or medical diagnosis of uncontrolled glaucoma (defined as IOP >25mmHg even with anti-glaucoma medication), advanced glaucoma resulting in a cup/disc ratio >0.8 in the study eye, or glaucoma filtration surgery in the study eye
* Serious complications following surgery in the study eye within 1 year
* Current or planned use of medications known to be toxic to the retina, lens, or optic nerve (e.g., deferoxamine, chloroquine/hydro chloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol)
* Medical history or condition: Uncontrolled diabetes mellitus, with glycosylated hemoglobin (HbA1c) > 10%, myocardial infarction or stroke within 12 months of screening, active bleeding disorder, major surgery within 1 month of screening or when planned within the study period, hepatic impairment, uncontrolled hypertension, other unstable or progressive cardiovascular, pulmonary, Parkinson, liver, or renal disease or cancer or dementia
* Previous treatment with intravenous bevacizumab or intravitreal ranibizumab, bevacizumab, aflibercept, pegaptanib in either of the eyes within four months prior to enrolment
* Previous treatment with verteporfin photodynamic therapy (PDT), thermal laser, transpupillary thermotherapy, intravitreal or protein kinase C inhibitors or other AMD therapy in the study eye within 3 months prior to randomization
* Previous treatment with intravitreal ocular or periocular steroids (e.g., triamcinolone, anecortave acetate) or peribulbar steroid in the study eye within past 3 months
* Concurrent use of systemic anti-VEGF agents
* Any ophthalmic device implantation within the previous 12 months
* Patients with a clinically significant abnormal screening hematology, blood chemistry, or urinalysis, unsuitable for study participation in the investigator's opinion
* Aspartate Transaminase (AST), Alanine Transaminase (ALT), alkaline phosphatase, Gamma-glutamyl Transferase (GGT), total bilirubin, direct bilirubin, indirect bilirubin, and LDH ≥ 2.0-fold the upper limit of normal at screening
* Patient with impaired renal function defined as calculated creatinine clearance (CLCr) <30mL/min

  * Males: CLCr = [140 - a(years)] x weight(kg)/ 72 x serum creatinine (mg/dL)
  * Females: CLCr = [140 - a(years)] x weight(kg) (x 0.85)/ 72 x serum creatinine (mg/dL)
* Significant alcohol or drug abuse within past 2 years per investigator judgement
* Previous participation in other trials for treatment of wAMD with systemic administration if washout period from last administration is shorter than 3 months
* Significant disease or other medical conditions (as determined by medical history, examination, and clinical investigations at screening) that may, in the opinion of the investigator result in the any of the following:

  * Put the patient at risk because of participation in the study,
  * Influence the results of the study,
  * Cause concern regarding the patient's ability to participate in the study
* Known hypersensitivity to fluorescein or any of the ingredients used in the study drug formulation, or any of the medications used during the study
* Active infectious conjunctivitis in either eye
* Women of childbearing potential who are lactating or who are pregnant as determined by serum pregnancy test at screening
* Women of childbearing potential must have agreed to use adequate birth control methods for the duration of the study
* Post-menopausal women should have documented last MC 2 years before study participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The percentage of occurrence of Adverse Events (AE) | Screening, Day 0, Day 28, Day 56 & Day 84
The number of Adverse Events (AE) that occurs | Screening, Day 0, Day 28, Day 56 & Day 84
Change in IOP with study drug compared to placebo | Screening, Day 0, Day 28, Day 56 & Day 84
  Mean change in intraocular pressure (IOP) with study drug compared to placebo from baseline to end of study
Change in intraocular inflammation with study drug compared to placebo | Screening, Day 0, Day 28, Day 56 & Day 84
  Mean change in intraocular inflammation with study drug compared to placebo from baseline to end of study
Incidence and severity of ocular and non-ocular adverse events of CG-P5 peptide eye drops and Placebo | Day 0, Day 28, Day 56 & Day 84
  Mean change in incidence and severity of ocular and non-ocular adverse events of CG-P5 peptide eye drops and Placebo with study drug compared to placebo from baseline to end of study

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) of study drug compared to Eylea® and placebo as measured by ≥15 Early ETDRS letter score at the end of 84 days | Screening, Day 0, Day 28, Day 56 & Day 84
Change in CNV area on fluorescence angiography with study drug compared to Eylea® and placebo on day 28, day 56 and day 84 | Day 28, Day 56 & Day 84
Mean decrease in central retinal thickness on SD-OCT with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Mean decrease in total macular volume on optical coherence tomography with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Proportion of patients with change in BCVA with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Number of patients with change in BCVA with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Proportion of patients with change in intraocular pressure (IOP) with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Number of patients with change in intraocular pressure (IOP) with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Proportion of patients with change in intraocular inflammation with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Number of patients with change in intraocular inflammation with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Proportion of patients with change in central retinal thickness with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Number of patients with change in central retinal thickness with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Proportion of patients with change in total macular volume with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Number of patients with change in total macular volume with study drug compared to Eylea® and placebo from baseline to end of study | Screening, Day 0, Day 28, Day 56 & Day 84
Change from Baseline in Choroidal Neovascularization (CNV) area as measured by Fluorescein Angiography (FA) over the study duration | Screening, Day 0, Day 28, Day 56 & Day 84
Change from Baseline in Central Subfield Thickness (CST) as measured by spectral domain optical coherence tomography (SD-OCT) over the study duration | Screening, Day 0, Day 28, Day 56 & Day 84
Area under the concentration-time curve from dosing (time 0) to time t [AUC(0-t)] | Day 0 & Day 84
  Pharmacokinetic profile of CG-P5 peptide eye drops measured by AUC(0-t)
Maximum Plasma Concentration [Cmax] | Day 0 & Day 84
  Pharmacokinetic profile of CG-P5 peptide eye drops measured by Cmax
Time of peak plasma concentration [Tmax] | Day 0 & Day 84
  Pharmacokinetic profile of CG-P5 peptide eye drops measured by Tmax
Half-life [t½] | Day 0 & Day 84
  Pharmacokinetic profile of CG-P5 peptide eye drops measured by t½

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yong Ji Chung, Study Director — Caregen Co. Ltd.
Locations (7):
- United States (7):
  - CBCC Global Research Site:005, Manchester, Connecticut
  - CBCC Global Research Site:006, Deerfield Beach, Florida
  - CBCC Global Research Site:001, Augusta, Georgia
  - CBCC Global Research Site:004, Carmel, Indiana
  - CBCC Global Research Site:003, Fargo, North Dakota
  - CBCC Global Research Site:002, Erie, Pennsylvania
  - CBCC Global Research Site:007, Philadelphia, Pennsylvania